CLINICAL TRIAL: NCT06193889
Title: KYSA-6: A Phase 2/3, Open-Label, Randomized, Controlled, Multicenter Study of KYV-101, an Autologous Fully Human Anti-CD19 Chimeric Antigen Receptor T-cell (CD19 CAR T) Therapy, Versus Ongoing Standard-Of-Care Immunosuppressive Therapy in Patients With Generalized Myasthenia Gravis
Brief Title: KYSA-6: A Study of Anti-CD19 Chimeric Antigen Receptor T-Cell Therapy, in Patients With Generalized Myasthenia Gravis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kyverna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KYSA-6; KYV101-006 (Other: Kyverna Therapeutics)
Record Dates: First submitted 2023-10-11; First posted 2024-01-05 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-09

CONDITIONS: Myasthenia Gravis; Generalized Myasthenia Gravis
Keywords: KYV-101; myasthenia gravis; autoimmune disease; anti-CD19 CAR-T Therapy; cellular therapy; MG; KYSA-6; KYV101-006
MeSH Terms: conditions — Myasthenia Gravis; Autoimmune Diseases | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- KYV-101 CAR-T cells with lymphodepletion conditioning (Experimental): Phase 2: Dosing with KYV-101 CAR-T cells
  Interventions: Drug: Standard lymphodepletion regimen; Biological: KYV-101
- KYV-101 Treatment (Experimental): Phase 3
  Interventions: Drug: Standard lymphodepletion regimen; Biological: KYV-101
- Standard of Care (Active Comparator): Phase 3 Optional crossover to receive KYV-101 Treatment after 24 weeks
  Interventions: Drug: Standard of Care Treatment; Drug: Standard lymphodepletion regimen; Biological: KYV-101

INTERVENTIONS:
Drug: Standard of Care Treatment — Standard of Care Medications Optional Crossover to receive KYV-101 treatment
  Arms: Standard of Care
Drug: Standard lymphodepletion regimen — Standard lymphodepletion regimen
  Other Names: Cyclophosphamide; Fludarabine
Biological: KYV-101 — Anti-CD19 CAR-T cell therapy

SUMMARY:
A Study of the Anti-CD 19 Chimeric Antigen Receptor T Cell Therapy for Patients with Myasthenia Gravis

DETAILED DESCRIPTION:
Myasthenia gravis (MG) is a chronic autoimmune disease that affects the neuromuscular junction and is characterized by muscle weakness. B cells play a role in MG, and the disease is characterized by the presence of autoantibodies such as anti-AChR and anti-MuSK antibodies. CD-19 target chimeric antigen receptor (CAR) T cells harness the ability of cytotoxic T cells to directly and specifically lyse target cells to effectively deplete both normal and autoreactive B cells in the circulation as well as impacted lymphoid and potentially non-lymphoid tissues. KYV-101, a fully human anti-CD19 CAR T-cell therapy, will be investigated in adult subjects with myasthenia gravis (MG).

ELIGIBILITY:
Key Inclusion Criteria

1. Presence of autoantibodies to AChR or MuSK at screening.
2. Myasthenia Gravis Foundation of America (MGFA) Class II-IV
3. MG-Activities of Daily Living (MG-ADL) total score of ≥6 at screening and confirmed at pre-dose baseline
4. QMG total score of ≥11 at screening an confirmed at pre-dose baseline
5. Failed treatment with 2 or more immunosuppressive/immunomodulatory therapies, or failed at least 1 immunosuppressive therapy and required chronic plasmapheresis, or IVIG (>4 times/year over ≥12 months) to control symptoms
6. On a stable dose of glucocorticoids and/or other immunotherapies for ≥1 month prior to screening. For patients treated with azathioprine, a stable dose for ≥2 months prior to screening is required
7. No change in dose of acetylcholinesterase inhibitors for ≥2 weeks prior to screening
8. No use of intravenous immune globulin (IVIG) or plasmapheresis (PLEX) within 4 weeks of screening or pre-dose baseline (unless this is part of their SOC treatment regimen)
9. No use of rituximab (or any other anti-CD20 or CD19 monoclonal antibody) within 12 weeks prior to screening
10. No use of FcRn inhibitors within 4 weeks prior to screening

Key Exclusion Criteria

1. Unable to washout or interrupt autoimmune disease therapy prior to apheresis
2. Co-occurring neurological autoimmune disease (ie, Lambert-Eaton Myasthenic Syndrome) or any disease affecting the neuromuscular junction or muscle causing weakness (eg, myositis, myopathy, motor neuropathy)
3. History of stroke (with residual sequalae and/or risk for recurrence), seizure (even if well controlled on antiepileptics), neurodegenerative disease, altered mental status (unexplained and/or recent/current), or uncontrolled/severe psychiatric disease
4. Any serious and/or uncontrolled medical condition that, in the investigator's judgment, would cause unacceptable safety risk, interfere with study procedures or results, or compromise compliance with the protocol, including but not limited to, clinically significant cardiac or pulmonary disease
5. History of primary immunodeficiency, organ or allogeneic bone marrow transplant, or splenectomy
6. Active, uncontrolled, viral, bacterial, or systemic fungal infection or recent history of repeated infections
7. Thymectomy <12 months of screening or planned during the study
8. Prior treatment with gene therapy product or cellular immunotherapy (eg, CAR T) requiring vector integration and directed at any target
9. Patients requiring chronic anticoagulation therapy that cannot be discontinued for medical procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) and laboratory abnormalities (Phase 2) | 2 years
Efficacy of KYV-101 via Myasthenia Gravis Activities of Daily Living (MG-ADL) change from baseline (Phase 2) | 24 weeks
Efficacy of KYV-101 via Myasthenia Gravis Activities of Daily Living (MG-ADL) change from baseline for KYV-101 Treatment Arm to Standard of Care Arm (Phase 3) | 24 weeks
Efficacy of KYV-101 via Quantitative Myasthenia Gravis (QMG) change from baseline for KYV-101 Treatment arm to Standard of Care arm | 24 weeks

SECONDARY OUTCOMES:
Efficacy of KYV-101 via Myasthenia Gravis Composite (MGC) score change from baseline for KYV-101 arm to Standard of Care arm (Phase 3) | 24 weeks
Efficacy of KYV-101 via Percent change from baseline in anti acetylcholine receptors (anti-AChR) antibody levels for KYV-101 Treatment arm to Standard of Care arm (Phase 3) | 24 weeks
Efficacy of KYV-101 via Percent change from baseline in anti muscle-specific tyrosine kinase (anti-MuSK) antibody levels for KYV-101 Treatment arm to Standard of Care arm (Phase 3) | 24 weeks
Efficacy of KYV-101 via Proportion of patients with a ≥3 point improvement from baseline in Myasthenia Gravis Activities of Daily Living (MG-ADL) for KYV-101 Treatment arm to Standard of Care arm (Phase 3) | 24 weeks
Efficacy of KYV-101 via Proportion of patients with minimal symptom expression (MSE) for KYV-101 Treatment arm to Standard of Care arm (Phase 3) | 24 weeks
Efficacy of KYV-101 via Myasthenia Gravis Quality of Life 15-item Scale (MG-QoL 15r) change from baseline for KYV-101 Treatment arm to Standard of Care arm (Phase 3) | 24 weeks
Incidence and severity of adverse events (AEs) and laboratory abnormalities (Phase 3) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Kyverna Therapeutics, Inc.
Locations (14):
- United States (7):
  - University of California, Irvine, Orange, California
  - Stanford University Medical Center, Palo Alto, California
  - University of Miami, Miami, Florida
  - Indiana University Health, Indianapolis, Indiana
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Houston Methodist Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
- Hospital Israelita Albert Einstein, São Paulo, Brazil
- Germany (6):
  - Charite- Universitätsklinikum Berlin, Berlin
  - Universitätsklinikum der Ruhr-Universität Bochum, Bochum
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochscule Hannover, Hanover
  - Friedrich-Schiller-Universität Jena, Jena
  - Universitätsklinik Magdeburg, Magdeburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gilhus NE, Tzartos S, Evoli A, Palace J, Burns TM, Verschuuren JJGM. Myasthenia gravis. Nat Rev Dis Primers. 2019 May 2;5(1):30. doi: 10.1038/s41572-019-0079-y. PMID 31048702